CLINICAL TRIAL: NCT02596672
Title: Promoting Walking in Older Adults Living in Independent Living Communities in Northern Ireland: A Feasibility Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Dr Mark Tully, Lecturer in Physical Activity and Public Health, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15.30
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Physical Activity; Aging; Health Behaviour; Social Isolation
Keywords: physical activity; older adults; retirement homes; walking; feasibility study
MeSH Terms: conditions — Motor Activity; Social Isolation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): They will complete a 12-week peer-led walking programme. Participants will be paired together as walking partners and will be given a pedometer and step count logs for self-monitoring. The walking co-ordinators will facilitate walking groups two times a week in the local areas, lasting for 30 minutes. The nature of the walks will be tailored to the participants stated preferences of types of activity. Participants will also receive local walking route maps. After 12 weeks, the formal peer-led component will finish and participants will be encouraged to continue walking with their walking partners other activity programmes organised in the fold in order to maintain activity levels.
  Interventions: Behavioral: The friendly walking group
- Control (No Intervention): Folds assigned to the control group will not receive any additional support to change their physical activity behaviour over the course of the intervention period.
  At the six-month data collection point they will be offered a referral to a local walking group in their area or advice on beginning a self-directed walking programme (similar to Public Health Agency www.choosetolivebetter.com/content/getting-active). They will be asked to complete outcome measures at baseline and follow up time-points. Post-study a sample of control participants will be asked to attend a focus group, exploring their views on social activity as form of physical activity for older adults in folds.

INTERVENTIONS:
Behavioral: The friendly walking group — A 12 week peer led walking group for adults and older adults (> 55 years) living in independent living communities in Northern Ireland. Designed to increase physical activity levels of inactive older adults and measure sustained changes in physical behaviour 6 months after the intervention ends.
  Arms: Intervention

SUMMARY:
The multi-level 12 week peer-led walking intervention incorporates aspects from all three levels of the ecological model (with the aim of producing sustained (>6months) physical activity behaviour change in older adults living in independent living communities.

DETAILED DESCRIPTION:
The proposed study is a cluster randomized controlled feasibility trial of a multi-level peer-led walking intervention. The socio-ecological model and social cognitive theory provides the framework that will help inform and test the feasibility of a multi-level peer-led walking intervention for inactive older adults living in independent living communities in Northern Ireland. The behaviour change techniques identified and extracted from a previous systematic review on the effectiveness of peer-led physical activity interventions helped guide the decision-making process of which behavior change strategies should be included in this study. The logic model helped inform the design and development of the 12 week peer-led walking programme.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over the age of 60 years recruited from fold housing associations, dependent on site; those receiving nursing care will not be included.
2. Inactive/not regularly walking (less than 30 minutes
3. Have the ability to read, write, understand and speak English.
4. Can walk freely without human assistance (residents will be included they use a walking stick/walking aid.)

Exclusion Criteria:

1. If they have fallen in the last 6 months
2. Have regular nursing assistance/care within the fold
3. Residents with dementia or other cognitive challenges will be excluded.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity (MVPA) | Baseline, 12 weeks and 6 months
  Changes from baseline MVPA as assessed by Actigraph accelerometer

SECONDARY OUTCOMES:
Quality of Life | Baseline, 12 weeks and 6 months
  To explore changes in health-related quality of life, a validated self-reported questionnaire EuroQol-5D will be completed by study participants.
Self-efficacy | Baseline, 12 weeks and 6 months
  Changes in self-efficacy will be measured using a short version of exercise behaviour self-confidence questionnaire.
Physical and Mental Health | Baseline, 12 weeks and 6 months
  Changes in other health-related and well-being outcomes will include completing the (7 item) Warwick-Edinburgh Mental Well-being score.
Social Engagement | Baseline, 12 weeks and 6 months
  Changes in social engagement will be measured using the Lubben social network scale

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Tully, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Centre for Public Health, Queen's University Belfast, Belfast, United Kingdom